CLINICAL TRIAL: NCT02791620
Title: The Efficacy of Nanofractional Radiofrequency Device in Arm Rejuvenation and Tightening : a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 256/59
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Skin Tightening and Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A nanofractional radiofrequency device (Experimental)
  Interventions: Device: a nanofractional radiofrequency device

INTERVENTIONS:
Device: a nanofractional radiofrequency device — A nanofractional radiofrequency device. noninvasive fractional radiofrequency device that provides ability to control and adjust the ratio of ablation and coagulation effect. Venus Viva, licensed by Health Canada, is cleared by the FDA for ablation and resurfacing dermatological procedures.
  Other Names: Venus Viva, Venus concept

SUMMARY:
The objective of this study is to evaluate arm rejuvenation and tightening with a nanofractional radiofrequency device, Venus viva, Venus concept, Toronto Canada. We recruit 20 subjects. All 20 subjects are treated with 3 sessions, 1 month interval with a nano fractional radiofrequency device on the inner upper arm. We evaluate skin tightening using %improvement of treated surface areas and skin elasticity using Dermalab the result at 3 months after the last treatment and clinical improvements evaluated by two board certified dermatologist (using compared photos between before treatment and 3 months after the last treatment).

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy female or male subjects, at least 30-60 years old of age 2. Subject who has BMI 18.50- 25 kg/m2 (as picture criteria above) 3. Subject has clinically evident moderate skin laxity with or without wrinkle on the upper arm 4. Subject has read and signed a written informed consent form.

Exclusion Criteria:

- 1. Patient with weight loss > 15% 2. Pregnancy or Lactation 3. History of pacemaker, defibrillator 4. History of laser resurfacing, prior radiofrequency, ultrasound or focused ultrasound on treatment areas within 1 year on the treatment area 5. History of Heat sensitivity, collagen vascular disorder disease including morphea, scleroderma, heat contact urticaria 6. History of medical illness that primary investigator thinks could interfere or influence the wound healing process 7. History of abnormal scars (keloid, hypertrophic scars) 8. History of skin cancer, radiation therapy or metal implants on treatment areas 9. Active local or systemic infection on treatment areas 10. Any other conditions that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

11. Subject is unable or unwilling to comply with the study requirements. 12. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Effects of arm rejuvenation and tightening | 12 weeks after the last treatment
  Determined by changing of the treated surface area (calculated from four-fixed tattoo points on the inner arm) surface area = length x width cm2

SECONDARY OUTCOMES:
Changing of skin laxity and elasticity | 12 weeks after the last treatment
  Evaluated by skin's viscoelastic properties using Dermalab, Courage Khazaka Electronic GmbH
Changing of skin wrinkles and laxity using photographs of subjects' baselines and 12 weeks after the last treatment by two independent board certified dermatologists | 12 weeks after the last treatment
  Determined by five point scale. (1) excellent improvement (>75%), (2) good improvement (50-75%), (3) fair improvement (25-50%), (4) some improvement (10-25%) and (5) little or no improvement (0-10%)
evaluate perceptions of treatment with a nano-fractional radiofrequency device | 12 weeks after the last treatment
  using five-point scale Five point scale evaluation: (1) excellent improvement (>75%), (2) good improvement (50-75%), (3) fair improvement (25-50%), (4) some improvement (10-25%) and (5) little or no improvement (0-10%)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsaie ML, Choudhary S, Leiva A, Nouri K. Nonablative radiofrequency for skin rejuvenation. Dermatol Surg. 2010 May;36(5):577-89. doi: 10.1111/j.1524-4725.2010.01510.x. Epub 2010 Apr 2. No abstract available. PMID 20384760
- [Background] Hruza G, Taub AF, Collier SL, Mulholland SR. Skin rejuvenation and wrinkle reduction using a fractional radiofrequency system. J Drugs Dermatol. 2009 Mar;8(3):259-65. PMID 19271373
- [Background] Hantash BM, Ubeid AA, Chang H, Kafi R, Renton B. Bipolar fractional radiofrequency treatment induces neoelastogenesis and neocollagenesis. Lasers Surg Med. 2009 Jan;41(1):1-9. doi: 10.1002/lsm.20731. PMID 19143021
- [Background] Sukal SA, Geronemus RG. Thermage: the nonablative radiofrequency for rejuvenation. Clin Dermatol. 2008 Nov-Dec;26(6):602-7. doi: 10.1016/j.clindermatol.2007.09.007. PMID 18940540
- [Background] Desai S. Nonsurgical Lifting and Tightening. Evidence-Based Procedural Dermatology: Springer; 2012. p. 287-300.